CLINICAL TRIAL: NCT06098703
Title: CARD (Comfort Ask Relax Distract) for Community-based Pharmacy Vaccinations
Brief Title: CARD for Community Pharmacy Vaccinations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Toronto (Other)
Collaborators: Public Health Agency of Canada (PHAC) (Other Government); Wholehealth Pharmacy Partners (Unknown)
Responsible Party: Principal Investigator, Anna Taddio, Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 43097
Record Dates: First submitted 2023-10-19; First posted 2023-10-24 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Vaccination Reaction; Vaccination Pain; Community Pharmacy
Keywords: Vaccination reaction; Vaccination experience

STUDY DESIGN:
Intervention Model Description: Cluster trial involving at least 24 community pharmacies allocated to CARD or control (standard care) in a 1:1 ratio. Eligible pharmacies belonging to Wholehealth Pharmacy Partners from across Ontario, Canada, will be included.
Who Masked: Participant, Outcomes Assessor
Masking Description: Vaccine recipients will not be aware of whether they are in the intervention or control group or the objective of the trial. Care providers who are trained in the intervention are aware of the group allocation. They will not communicate with care providers not trained in the intervention. Care providers that are in the intervention pharmacies will not deliver care to participants in the control pharmacies and care providers in the control pharmacies will not deliver care in the intervention pharmacies. Vaccine recipients are rating the primary outcome.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CARD (multi-faceted intervention) (Experimental): CARD will be integrated in the pharmacy vaccination process. This includes education, environment (e.g., clinic spaces), engagement (interactions), and evaluation (surveys/feedback).
  Interventions: Behavioral: CARD (Comfort Ask Relax Distract)
- Control (standard care) (No Intervention): There are no specific procedures being undertaken to plan or execute vaccine clinics. Usual practices will be instituted by participating pharmacies.

INTERVENTIONS:
Behavioral: CARD (Comfort Ask Relax Distract) — CARD is a vaccine delivery framework/protocol to plan and deliver vaccinations
  Arms: CARD (multi-faceted intervention)

SUMMARY:
To integrate CARD in community pharmacy-led vaccinations and document impact on vaccine clients and pharmacy staff.

DETAILED DESCRIPTION:
It is estimated that 1 out of 5 children and adults are not vaccinated because of concerns about pain and fear. The CARD (Comfort Ask Relax Distract) system is a new vaccine delivery system proven to reduce pain, fear and immunization stress-related responses. Improving the vaccination experiences of patients can improve attitudes about vaccination and increase vaccine acceptance.

The objective of this cluster randomized trial is to evaluate scaling of CARD across community pharmacies on patients vaccination symptoms, beliefs and attitudes and pharmacy staff beliefs and attitudes.

ELIGIBILITY:
Inclusion Criteria:

* vaccine clients being vaccinated in community pharmacies participating in the project
* pharmacy staff in community pharmacies participating in the project

Exclusion Criteria:

* unable to understand and read English

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Experience with vaccination | within 15 minutes after vaccination
  Vaccine client self-reported experience with vaccination (better or not)

SECONDARY OUTCOMES:
Fear | within 15 minutes after vaccination
  Vaccine client self-reported fear during vaccination (0-10)
Pain | within 15 minutes after vaccination
  Vaccine client self-reported pain during vaccination (0-10)
Dizziness | within 15 minutes after vaccination
  Vaccine client self-reported dizziness during vaccination (0-10)
Fainting | within 15 minutes after vaccination
  Fainting during/after vaccination (yes/no)
Utilization of coping strategies during vaccination | within 5 minutes of vaccination
  Use of individual coping strategies during vaccination (e.g., distraction, support person) (yes/no)
CARD satisfaction survey | within 15 minutes of vaccination
  Vaccine client self-reported satisfaction with CARD (e.g., helpfulness, willingness to use again, willingness to return for next vaccination, vaccination decision-making, as applicable), responses reported for individual items
Implementation success of CARD | within 3 months of vaccination clinics
  Perceptions of implementation success of CARD program delivery as reported by CARD implementers (primary targets) using CARD Global Impression Checklist, individual questions (5-point Likert Scale higher number represents better outcome); responses reported for individual items. This information is supplemented with focus group information and study notes.
Attitudes about vaccination | within 3 months of vaccination clinics
  Perceptions of CARD and non-CARD implementers using CARD Attitudes survey, individual questions (5-point Likert Scale higher number represents better outcome); responses reported for individual items. This information is supplemented with focus group information and study notes.
Vaccination behaviours | within 3 months of vaccination clinics
  Self-reported vaccine behaviours of immunizers using CARD Behaviour Survey, individual questions (rank as whether behaviours are done or not); responses reported for individual items. Includes CARD and non-CARD implementers.
Vaccine interaction survey | within 5 minutes of vaccination
  Perceptions of CARD and non-CARD immunizers about vaccination interaction [duration, satisfaction, CARD usefulness (intervention group only)]; responses reported for individual items.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Taddio, PhD, Principal Investigator — University of Toronto
Locations (1):
- Anna Taddio, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
We do not have permission to share this information.

REFERENCES:
- [Derived] Taddio A, Morrison J, Logeman C, Gudzak V, Bucci LM, McMurtry CM, Yang M, Folinas M, Moineddin R, MacDonald NE. CARD (Comfort Ask Relax Distract) and community pharmacy vaccinations: Evaluation of effectiveness outcomes from a cluster randomized trial. Hum Vaccin Immunother. 2025 Dec;21(1):2488064. doi: 10.1080/21645515.2025.2488064. Epub 2025 Aug 6. PMID 40768541
- [Derived] Taddio A, Morrison J, Logeman C, Gudzak V, Bucci LM, McMurtry CM, Yang M, Folinas M, Moineddin R, MacDonald NE. CARD (Comfort Ask Relax Distract) and community pharmacy vaccinations: Evaluation of implementation outcomes from a cluster randomized trial. Hum Vaccin Immunother. 2025 Dec;21(1):2503524. doi: 10.1080/21645515.2025.2503524. Epub 2025 May 15. PMID 40371950